CLINICAL TRIAL: NCT04814680
Title: A Non-Interventional Pilot Study to Evaluate A Machine-Learning Algorithm for Prediction of Blood Pressure, Glycated Haemoglobin and Estimated Glomerular Filtration Rate From Digital Retinal Images
Brief Title: Machine-Learning Algorithm for Prediction of Blood Pressure, Glycated Haemoglobin and Estimated Glomerular Filtration Rate
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D9080C00001
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Prediction of Blood Pressure, Glycated Haemoglobin and Estimated Glomerular Filtration Rate From Digital Retinal Images
Keywords: - Machine learning; retinal images; blood pressure; glycated haemoglobin; glomerular filtration rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional pilot study with the following objectives:

* Establish scalable methodology for collection of retinal images, blood pressure (BP) and laboratory-based assessments
* Compare the results of a machine-learning algorithm in predicting BP, glycated haemoglobin (HbA1c) and estimated glomerular filtration rate (eGFR) from digital retinal images with clinical and laboratory-based measures
* Determine the required sample size needed to support a future study to fully validate the machine-learning algorithm

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 35 years of age, at the time of signing the informed consent.
* With or without DM (at least 50% of participants will have an HbA1c ≥ 6.5%* and/or a known diagnosis of DM)
* Male or female (at least 40% of participants must be male, and at least 40% must be female)
* Capable of giving signed informed consent as described in Appendix A

Exclusion Criteria:

* As judged by the investigator, any evidence of a medical condition which in the investigator's opinion makes it undesirable for the participant to participate in the study for example, but not limited to, if a participant is critically unwell or requiring ongoing emergency treatment
* Any known eye condition that may preclude clear imaging of the retina for example; cataracts
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
* Previous enrolment in the present study with the exception of roll-in participants who may be re-screened and re-enrolled.

Ages: 35 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have to be more than 35 years, able to provide written consent and meet the following inclusion criteria:
  * With or without DM (at least 50% of participants will have an HbA1c ≥ 6.5%* and/or a known diagnosis of DM)
  * Male or female (at least 40% of participants must be male, and at least 40% must be female)
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
To assess successful use of methodology for retinal image acquisition, BP (ABPM or manual), HbA1C (laboratory based or point of care test) and e-GFR measurement. | up to 66 day
  Proportion of participants with completed study procedures and interpretable results including both retinal images, systolic and diastolic BP (ABPM or manual), HbA1c (laboratory based or point of care test) and eGFR at Visit 1

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9080C00001&attachmentIdentifier=5cdc1cb2-be84-4f97-ac61-b2cb6257f5b0&fileName=d9080c00001-clinical-study-report_synopsis_Redacted.pdf&versionIdentifier=